CLINICAL TRIAL: NCT01158157
Title: Vaccinia Vaccine (ACAM2000) for the Production of Vaccinia Immune Globulin Intravenous (VIGIV)
Brief Title: VA-006 Vaccinia Vaccine (ACAM2000) for the Production of VIGIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VA-006
Record Dates: First submitted 2010-07-05; First posted 2010-07-08 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Smallpox Vaccine Adverse Reaction
MeSH Terms: interventions — ACAM2000

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vaccination (Other): This study was a single arm study. All eligible subjects received ACAM2000.
  Interventions: Biological: ACAM2000

INTERVENTIONS:
Biological: ACAM2000 — Percutaneous administration of a droplet (2.5µg) of ACAM2000 using a bifurcated needle.

SUMMARY:
The purpose of this study is to vaccinate plasma donors with ACAM2000 smallpox vaccine for collection of plasma to be used in the manufacturing of Vaccinia Immune Globulin Intravenous (VIGIV).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Age 18 - 65 years.
* Normal and healthy as determined by medical history, physical exam, vital signs and clinical laboratory tests at screening visit.
* Subject must meet all required subject suitability criteria that pertain to normal Source Plasma donors.
* Subject must have been previously immunized for smallpox, at ≥1 year prior to commencement of screening assessments for the VA-006 trial, and vaccination history must be confirmed by oral or written history AND the presence of a visible pathognomonic smallpox vaccination scar.
* Female subjects of childbearing potential must use at least one of the following means of birth control documented by a physician's letter:

  * Surgical sterilization
  * Hormonal (oral/injectable/implant) for at least 30 days prior to vaccination
  * Intrauterine device (IUD) inserted at least 7 days prior to vaccination.
* Female subjects who are not using one of the methods of birth control listed above must be documented as postmenopausal, which is defined as not having a menstrual period for longer than 12 months and having a serum follicle-stimulating hormone (FSH) level ≥ 40 mIU/mL.

Exclusion Criteria:

* History of severe adverse event(s) from previous participation in the VA-001 or VA-005 trials or any other smallpox vaccination program/study.
* Subject, household contact, or other close/intimate contact:

  * with eczema, history of eczema, exfoliative skin conditions, wounds, burns, or other skin conditions at the Investigator's discretion.
  * with a history of immunodeficiencies (see section 7.1.2 of the protocol).
  * who received radiotherapy or chemotherapy, adrenocorticotropic hormone (ACTH), corticosteroids, or immunosuppressive drugs.
  * with eye disease treated with topical steroids.
  * with known or suspected disorders of immunoglobulin synthesis.
  * with leukemia, lymphomas of any type, melanoma, or other malignant neoplasms affecting the bone marrow or lymphatic systems.
  * with a history of adverse reactions to smallpox (vaccinia) vaccine.
  * has recently been diagnosed with cancer and who will be undergoing chemotherapy or radiation therapy during the vaccination healing time.
  * is a transplant recipient (except for corneal transplant).
  * is pregnant, planning pregnancy or breast feeding (female subjects must have negative serum pregnancy test at screening and negative urine pregnancy test prior to vaccination).
* Household or other close/intimate contact(s) under the age of 12 months.
* History of allergies to latex, phenol, any of the antibiotics listed in the vaccine content, or any other component of ACAM2000 or its diluent
* Severely or morbidly obese or higher obesity classification (BMI ≥ 35).
* Subjects with abnormal EKG and/or cardiac Troponin levels at screening.
* Subjects with cancer or kidney disease (except kidney stones).
* Subject has 3 or more of the following risk factors:

  * High blood pressure diagnosed by a doctor
  * High blood cholesterol diagnosed by a doctor
  * Diabetes or high blood sugar diagnosed by a doctor
  * A first degree relative (for example, mother, father, brother, sister) who had a heart condition before the age of 50
  * Currently smokes cigarettes
* Cardiovascular disease or heart condition diagnosed by a doctor at any time in the past, with or without symptoms, including:

  * Arrhythmia
  * Syncope
  * Previous myocardial infarction
  * Angina
  * Coronary artery disease
  * Congestive heart failure
  * Cardiomyopathy
  * Stroke or transient ischemic attack
  * Chest pain or shortness of breath with activity (such as walking up stairs)
  * Other heart conditions being treated by a physician.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-09-13 (Actual); Primary Completion 2012-02-14 (Actual); Study Completion 2012-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Brown, MD, Principal Investigator — Cangene Plasma Resources, Mid-Florida
Locations (1):
- Cangene Plasma Resources, Mid-Florida, Altamonte Springs, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Russell PK. Vaccines in civilian defense against bioterrorism. Emerg Infect Dis. 1999 Jul-Aug;5(4):531-3. doi: 10.3201/eid0504.990413. No abstract available. PMID 10458959
- See also: World Health Organization. Declaration of global eradication of smallpox. Wkly. Epidemiol. Rec., 55:145-152, 1980. — http://whqlibdoc.who.int/wer/WHO_WER_1980/WER1980_55_145-152%20(N%C2%B020).pdf
- See also: Centers for Disease Control and Prevention (CDC). Public Health Service recommendations on smallpox vaccination. MMWR, 20:339, 1971. — http://www.cdc.gov/mmwr/
- See also: CDC. Recommendation of the Immunization Practices Advisory Committee (ACIP). Smallpox vaccination of hospital and health personnel. MMWR, 25:9, 1976. — http://www.cdc.gov/mmwr/
- See also: CDC. Smallpox vaccine no longer available for civilians-United States. MMWR, 32:387, 1983. — http://www.cdc.gov/mmwr/
- See also: CDC. Vaccinia (smallpox) vaccine recommendations of the Immunization Practices Advisory Committee (ACIP). MMWR, 40:1-10, 1991. — http://www.cdc.gov/mmwr/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vaccination
Started | 25 (61 subjects screened; 25 subjects were vaccinated; 36 subjects were not eligible.)
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: A total of 61 subjects were screened for VA-006 study; 25 subjects satisfied the eligibility criteria and were percutaneously administered ACAM2000 vaccine, while 36 subjects were not eligible for the study and were not administered ACAM2000.
Arm/Group | Vaccination
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 25
Age [Mean (Standard Deviation); unit: years] | 47 (9.1)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Adverse Events Related to ACAM2000 Vaccine Administration
Time Frame: Days 0 to 90 post-vaccination
Population: Post-vaccination adverse events were assessed in the safety population.
Measure: Number; unit: percentage of participants
Groups:
- ACAM200 Vaccination Dose: Participants received a single percutaneous administration of a droplet (2.5 μL) of the ACAM2000 smallpox vaccine using a bifurcated needle on Day 0.
Arm/Group | ACAM200 Vaccination Dose
Number analyzed (Participants) | 25
percentage of participants
  Vaccination complications | 52
  Headache | 8
  injection site scab | 4

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Description: AE: Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Arm/Group | ACAM200 Vaccination Dose
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 15/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACAM200 Vaccination Dose (N=25)
Injection site scab (General disorders) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 13 (14)
Headache (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes